CLINICAL TRIAL: NCT01965522
Title: Anti-proliferative Effects of Vitamin D and Melatonin in Breast Cancer
Acronym: MELO-D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Juravinski Cancer Center (Other)
Responsible Party: Principal Investigator, Punam Rana, Principal Investigator, Juravinski Cancer Center
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MELO-D; NCT02288806 (obsolete NCT alias)
Record Dates: First submitted 2013-10-11; First posted 2013-10-18 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Early Stage Breast Cancer
Keywords: Breast cancer; melatonin; vitamin d; ki67
MeSH Terms: conditions — Breast Neoplasms | interventions — Melatonin; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Melatonin and Vitamin D (Experimental)
  Interventions: Drug: Melatonin; Drug: Vitamin D
- Placebo and Vitamin D (Experimental)
  Interventions: Drug: Vitamin D; Drug: Placebo (melatonin)
- Melatonin and Placebo (Experimental)
  Interventions: Drug: Melatonin; Drug: Placebo (vitamin D)
- Placebo and Placebo (Placebo Comparator)
  Interventions: Drug: Placebo (melatonin); Drug: Placebo (vitamin D)

INTERVENTIONS:
Drug: Melatonin — Melatonin 20mg taken orally once daily. This is in the form of one capsule which contains two pills of melatonin, 10 mg each.
  Arms: Melatonin and Placebo; Melatonin and Vitamin D
Drug: Vitamin D — Vitamin D 2000 IU taken orally once daily. This is in the form of one capsule which contains two pills of vitamin D, 1000 IU each.
  Arms: Melatonin and Vitamin D; Placebo and Vitamin D
Drug: Placebo (melatonin) — Overencapsulated placebo capsule which contains an inert substance. The capsule appears identical to the capsule which contains melatonin tablets.
  Arms: Placebo and Placebo; Placebo and Vitamin D
Drug: Placebo (vitamin D) — Overencapsulated placebo capsule which contains an inert substance. The capsule appears identical to the capsule which contains vitamin D tablets.
  Arms: Melatonin and Placebo; Placebo and Placebo

SUMMARY:
Investigators plan to carry out a study to investigate two different pills, Vitamin D and melatonin, and whether they can reduce the spread of cancer cells in the tumors of women with breast cancer. These pills are inexpensive and have very few side effects. A large number of studies using cell cultures and animals have shown that both vitamin D and melatonin can help destroy breast cancer cells. However thoughtful and well-designed studies are necessary on humans to see if they can decrease the spread of breast cancer, and possibly even prevent breast cancer. The proposed study aims to understand the anti-cancer activity of vitamin D and melatonin. This knowledge will assist in creating efficient cancer prevention strategies for Canadians. This study will include women with breast cancer who are being planned for surgery, and will assess whether treatment with vitamin D (dose of 2000 IU per day) in a group of 36 women, or melatonin (dose of 20mg per day) in another group of 36 women, or both pills together in yet another group of 36 women, reduces the spread of cancer cells when compared to a fourth group of 36 women who are treated with sugar pills. To do this we will measure a substance in the blood called Ki67, which provides information about the spread of cancer. Investigators will compare the Ki67 levels in the 4 groups, and all women will receive identical appearing pills so they will not know which treatment they received.

ELIGIBILITY:
Inclusion Criteria:

* Woman with histologically confirmed invasive breast cancer (ductal, lobular, or mixed)
* Planned to undergo definitive surgery, either lumpectomy or mastectomy in 3 or more weeks

Exclusion Criteria:

* Less than 18 years of age
* Stage IIIB or IV disease
* Inoperable locally advanced or metastatic breast cancer
* Neoadjuvant chemotherapy is intended
* Currently taking vitamin D supplements
* Currently taking melatonin supplements
* Previously taking vitamin D or melatonin supplements within the last 3 months
* Currently taking a multivitamin and not willing to discontinue for the duration of the study
* Hyperparathyroid disease or other calcium disturbance in the past five years
* Active renal stones in the last six months
* Renal failure (creatinine > 190 mmol/L)
* Hypercalcemia (serum calcium > 2.6 mmol/L)
* Known pregnancy
* Participation in another clinical trial where the patient receives any other investigational product
* Unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-10; Primary Completion 2016-08 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Ki67 | From time of initial biopsy to the final surgery, which is on average 4 weeks
  The primary outcome is the difference in proliferation rate of Ki67 in the tumour (expressed as the percentage of tumour cells expressing Ki67). Ki67 will be measured on the original core biopsy (pre-treatment) and on the lumpectomy/mastectomy specimen (post-treatment).

SECONDARY OUTCOMES:
microRNA | At the time of surgery compared to time of biopsy, which is on average 4 weeks
  Change in serum profile of microRNA at the time of surgery (lumpectomy or mastectomy, post-treatment) will be compared to the time of initial biopsy (pre-treatment).

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - St Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Juravinski Cancer Center, Hamilton, Ontario